CLINICAL TRIAL: NCT00002119
Title: A Phase I/II Clinical Study of WF 10 IV Solution ( TCDO ) in Patients With HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxo Chemie GmbH (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 222A; WF10-92-US-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex

INTERVENTIONS:
Drug: WF10

SUMMARY:
To evaluate the clinical toxicity, safety, and MTD of WF 10 ( TCDO ) intravenous solution administered to patients with HIV infection. To evaluate the potential anti-HIV activity of TCDO.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine (300 mg monthly) as prophylaxis for PCP only in patients with CD4 count <= 200 cells/mm3.

Allowed:

* PCP prophylaxis with aerosolized pentamidine in patients with CD4 count > 200 cells/mm3, only at the discretion of the treating physician.

Patients must have:

* HIV positivity.
* Absolute CD4 count of 150 - 500 cells/mm3.
* At least 6 months of prior zidovudine therapy.
* No active opportunistic infection requiring ongoing therapy.
* Life expectancy of at least 6 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Neoplasm other than basal cell carcinoma of the skin.
* Clinically significant cardiac disease.
* Abnormal neurological status by a standardized assessment including strength, reflex testing, and sensory testing.
* Unwilling to comply with protocol requirements.

Patients with the following prior conditions are excluded:

History of myocardial infarction or arrhythmias.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Antiretroviral agent or interferon.
* Systemic biologic response modifiers, corticosteroids, cytotoxic chemotherapeutic agents, or other drugs that can cause neutropenia or significant nephrotoxicity.
* Rifampin or rifampin derivatives.
* Systemic anti-infectives.

Required:

* At least 6 months of prior zidovudine. Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Oncol Med Associates, Houston, Texas, United States

REFERENCES:
- [Background] Busch HW, Christensen S, Reichelt D, Jahn S, Zidek W. Treatment of HIV-infected patients with advanced symptomatic disease with WF10 solution (TCDO). Int Conf AIDS. 1994 Aug 7-12;10(1):204 (abstract no PB0245)
- [Background] Kahn JO, McGrath MS, Ching OM, Kuhne FW. A single center, phase 2 study evaluating the effects of WF10. Int Conf AIDS. 1998;12:349 (abstract no 22423)
- [Background] Raffanti SP, Schaffner W, Federspiel CF, Blackwell RB, Ching OA, Kuhne FW. Randomized, double-blind, placebo-controlled trial of the immune modulator WF10 in patients with advanced AIDS. Infection. 1998 Jul-Aug;26(4):202-7. doi: 10.1007/BF02962364. PMID 9717676